CLINICAL TRIAL: NCT05638698
Title: Phase II Randomized Trial Combining Tg01 Vaccine / Qs-21 Stimulon™ With Or Without Balstilimab As Maintenance Therapy Following Adjuvant Chemotherapy In Patients With Resected Pancreatic Cancer(TESLA)
Brief Title: Tg01 Vaccine / Qs-21 Stimulon™ With Or Without Balstilimab As Maintenance Therapy Following Adjuvant Chemotherapy In Patients With Resected Pancreatic Cancer
Acronym: TESLA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Targovax ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00149222
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — saponin QA-21V1; balstilimab

STUDY DESIGN:
Intervention Model Description: This is a two arm, open-label, phase II randomized trial of TG01 vaccine and QS- 21 (vaccine arm) or TG01 vaccine and QS-21 plus Balstilimab (Vaccine + PD1i arm) in patients with surgically resected Stage 1-3 RAS mutant pancreatic cancer who have positive circulating tumor DNA (ctDNA+) in the blood despite prior standard therapy including chemotherapy/radiation therapy where applicable; no evidence of disease by imaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TG01/QS-21 (Vaccine arm) (Experimental): TG01 is mixed with adjuvant QS-21 and given subcutaneously. After six administrations given once every two weeks of TG01 vaccine (+adjuvant QS-21) over 12 weeks during weeks 1,3,5,7,9,11, [priming/booster phase]), the treatment will then switch to a maintenance phase of TG01 vaccine (+adjuvant QS-21) once every 8 weeks for up to 51 weeks: The maintenance treatments will occur during weeks 19, 27, 35, 43, and 51. Maintenance treatments will end on week 51 or at the time of disease recurrence; whichever is the earliest.
  Interventions: Biological: TG01 Vaccine; Drug: QS-21
- TG01/QS-21 + Balstilimab (Vaccine + PD-1 arm) (Experimental): TG01 is mixed with adjuvant QS-21 and given subcutaneously. Balstilimab is given intra-venously as infusion and begins week 3, then given every 2 weeks for up to 51 weeks. After six administrations given once every two weeks of TG01 vaccine (+adjuvant QS-21) over 12 weeks during weeks 1,3,5,7,9,11, [priming/booster phase]), the treatment will then switch to a maintenance phase of TG01 vaccine (+adjuvant QS-21) given once every 8 weeks for up to 51 weeks: The maintenance treatments will occur during weeks 19, 27, 35, 43, and 51. Maintenance treatments will end on week 51 or at the time of disease recurrence; whichever is the earliest.
  Interventions: Biological: TG01 Vaccine; Drug: QS-21; Drug: Balstilimab

INTERVENTIONS:
Biological: TG01 Vaccine — used to assess molecular disease control rate when combined with other interventional methods.
Drug: QS-21 — used to assess molecular disease control rate when combined with other interventional methods.
Drug: Balstilimab — used to assess molecular disease control rate when combined with other interventional methods.
  Arms: TG01/QS-21 + Balstilimab (Vaccine + PD-1 arm)

SUMMARY:
Researchers want to discover if the new drug "TG01" will work with participants' bodies to help their immune system attack any cancer cells that might still be in the blood stream after surgery for pancreatic cancer.

The researchers will also investigate whether or not "TG01" combined with the other study drug, "Balstilimab", will show even greater efficacy.

TG01 and Balstilimab are both experimental treatments and are not approved by the US Food and Drug Administration (FDA) as treatment in the United States, or elsewhere, for pancreatic cancer or any other type of cancer.

Balstilimab has been studied in other cancers and has shown signs of efficacy. Another drug will be used in this study called "QS-21". It is not intended to treat any disease but is used in this study to improve the action of the study drug TG01.

QS-21 has been approved by the US Food and Drug Administration (FDA) to be mixed with a vaccine used to prevent shingles. It has not been approved to be mixed with the study drug, TG01.

Participants will undergo eligibility screening, weekly visits during treatment when receiving the study drug or study drug combination, two safety follow-up visits, at about 30 and 90 days after the last dose of study treatment, and long term follow up for about 12 months after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 18 years
* ECOG Performance Status 0 - 1 within 28 days prior to registration (Appendix A)
* Surgically resected stage I/II/III Pancreatic Cancer
* Life expectancy of at least 6 months
* Screening tumor tissue positive or known pathogenic or likely pathogenic RAS mutation resulting in amino acid substitution in codon 12A, 12C, 12D, 12R, 12S or 13D . Mutations must be considered pathogenic or likely pathogenic by a reference database such as ClinVar or OncoKb.org.(https://www.ncbi.nlm.nih.gov/clinvar/variation;https://www.oncoKb.org). Local RAS test results are acceptable and central confirmation is not required prior to treatment.
* No evidence of recurrent cancer on screening imaging studies
* Positive for Minimal Residual Disease (MRD) as assessed by Signatera circulating tumor DNA (ctDNA) despite prior standard therapy including surgery and chemotherapy/radiation therapy where applicable
* Prior cancer treatment must be completed at least 14 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiating treatment. See also section with title CHILD BEARING POTENTIAL /PREGNANCY
* Adequate organ function, measured within 28 days prior to enrollment and defined as follows:

  * Hgb ≥ 8g/dL
  * Creatine clearance ≥ 50ml/min (measured or calculated by the Cockroft-Gault method)
  * Leukocytes >1.5K/UL
  * Absolute Neutrophil Count >1.5K/UL NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
  * Platelets >100K/UL
  * Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN
  * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
  * Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 30 days after the last dose of TG01/QS-21 immunotherapy and 90 days after the last dose of Balstilimab.

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Is pregnant, planning pregnancy, or breastfeeding
* Has a known allergic reaction to any excipient contained in the study drug formulation
* Has received an investigational drug within 4 weeks prior to study drug administration
* Is currently receiving any agent with a known effect on the immune system, unless at dose levels that are not clinically immunosuppressive (e.g. Prednisone at 10 mg/day or less, or as inhaled steroid at doses used for the treatment of asthma
* Has any other serious illnesses or medical conditions such as, but not limited to:

  1. Any uncontrolled infection
  2. Uncontrolled cardiac failure classification New York Heart Association (NYHA) III or IV
  3. Uncontrolled systemic and gastro-intestinal inflammatory conditions
  4. Inadequate bone marrow function with suspected inability to mount an immune response to vaccination
* Severe intercurrent disease which might affect immunocompetence
* Unacceptable values of the hematological or chemical tests (in relation to the ability to generate an immune response), as judged by the investigator
* Active or prior documented autoimmune disease within the past 2 years. Note: subjects with vitiligo, Grave's disease, psoriasis not requiring systemic treatment or hypothyroidism (i.e.

following Hashimoto syndrome) stable on hormone replacement are not excluded.

* Active or prior documented inflammatory bowel disease (i.e. ulcerative colitis)
* History of adverse reactions to peptide vaccines
* Positive tests for human immunodeficiency virus (HIV) or hepatitis B or C infection
* Planning to receive yellow fever or other live (attenuated) vaccines during the course of the study.
* Have any other active malignancies (except for adequately treated carcinoma of the cervix or basal or squamous cell skin cancer) which in the opinion of the investigator is likely to require treatment within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Molecular disease control rate | 6 months
  To assess 6-month molecular disease control rate in each cohort as defined by ctDNA stability, decrease or clearance.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  To assess safety of TG01/QS-21 safety with or without Balstilimab using CTCAE version 5.0
Disease free survival rate | 12 months
  To assess 6- month and 12-month Disease free survival rate in each cohort
Complete molecular response rate | 6 months
  To assess complete molecular response rate in each cohort as defined by ctDNA clearance
Correlation between molecular response and disease free survival | 6 months
  To assess the correlation between the depth of molecular response to disease free survival in each cohort

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, Principal Investigator — The University of Kansas Cancer Center
Locations (5):
- United States (5):
  - University of Kansas Cancer Center - Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No